CLINICAL TRIAL: NCT05999123
Title: Study for the Development of Biometrics-informed Menstrual Cycle Algorithms
Brief Title: Menstrual Cycle Study
Status: Completed | Type: Observational
Sponsor: Fitbit LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-FH-001
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-09

CONDITIONS: Menstruation; Ovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Up to 150 participants will be enrolled at one or more clinical research sites in the United States. Participants will be healthy, menstruating individuals between 18 to 42 years of age who meet all eligibility criteria.

SUMMARY:
A data collection study to develop algorithms to estimate menstrual cycle phases.

ELIGIBILITY:
Inclusion:

* Adults who are between 18 - 42 years old at enrollment and menstruate
* Capable of giving informed consent in Spanish or English
* Menstrual cycle lengths between 21- 45 days
* Have tracked menstruation for at least 3 menstrual cycles out of the prior 6 months
* Willing to wear a wrist-worn wearable device continuously for 6 months
* Willing to use an ovulation predictor kit for 6 months
* Willing to report vaccine history
* Owns a smartphone compatible with the study and has access to wi-fi

Exclusion:

* A citizen of the European Union or United Kingdom
* Trying to conceive during the six-month study period
* Have used specific forms of birth control in the 3 months prior to the study or planning on using specific birth control methods during the study duration
* Participant has undergone hormonal treatment in the past 3 months or planning to do so during the study
* Known history of health-related issues that affect their menstrual cycle, history of pelvic radiation, vasomotor symptoms, endometriosis, fibroids, polyps, ovarian cysts or known history of health-related issues that affect the physiology
* Currently (or within the past 3 months) engaged in health impacting behaviors
* Have been breastfeeding or pregnant in the past 6 months prior to the study
* On medications or taking substances that could affect their menstrual cycle or physiology
* Travel frequently such as crossing more than two time zones at least once every 2 weeks
* Have a known sleeping disorder or consistently work night shifts

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, menstruating individuals between 18 to 42 years of age who meet eligibility criteria from one or more clinical research sites in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Ovulation Day Estimation | 6 months
  The algorithm's estimated ovulation day compared to the reference urinary ovulation predictor kits (OPK).

SECONDARY OUTCOMES:
Menstruation Day Estimation | 6 months
  The algorithm's estimated menstruation date(s) compared to participants' self-reported menstruation date(s).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Johnson, DO, Principal Investigator — Artemis Institute for Clinical Research
Locations (1):
- Artemis Headlands LLC (Artemis Institute for Clinical Research), San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No